CLINICAL TRIAL: NCT00993941
Title: Evaluation the Efficacy and Safety of Autologous Bone Marrow Mesenchymal Stem Cells (MSCs) Transplantation in Patients With Early and Middle Stage of Liver Cirrhosis
Brief Title: Bone Mesenchymal Stem Cell (BMSC) Transplantation in Liver Cirrhosis Via Portal Vein
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Lin Bingliang, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-Bingliang
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2009-10

CONDITIONS: Liver Cirrhosis
Keywords: BMSC; Stem cells; Liver cirrhosis; Transplantation
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A(conserved therapy ) (Active Comparator): Thirty of the enrolled patients were randomly assigned to Group A were received comprehensive treatment including antiviral drugs, lowering aminotransferase and jaundice medicine.
  Interventions: Drug: Conserved therapy
- Group B (BMSC Transplantion) (Experimental): Thirty of the enrolled patients were randomly assigned to Group B were received comprehensive treatment including antiviral drugs, lowering aminotransferase and jaundice medicine, as well as Bone Mesenchymal Stem Cells(BMSC) transplantation via portal vein.
  Interventions: Procedure: Autologous BMSCs transplantation

INTERVENTIONS:
Procedure: Autologous BMSCs transplantation — 10 ml autologous BMSCs(7~8log10 cells/ml) were infused to patients using interventional method via portal vein as well as conserved therapy for group B.
  Arms: Group B (BMSC Transplantion)
Drug: Conserved therapy — Oral or intravenous administration
  Arms: Group A(conserved therapy )

SUMMARY:
The objective of this study is to evaluate the therapeutic efficacy of autologous bone marrow mesenchymal stem cells (BMSCs) transplantation via portal vein in patients with early and middle stage of liver cirrhosis on the basis of HBV infection. The evaluation of the efficacy includes the level of serum alanine aminotransferase (ALT), aspartate aminotransferase(AST), total bilirubin (TB),prothrombin time (PT), albumin (ALB), prealbumin(PA), precollagenⅢ(PCⅢ), collagenⅣ(Ⅳ-C), laminin(LN), hyaluronidase(HN), liver histological improvement before and 1 week to 1 year after transplantation. Child-Pugh scores and clinical symptoms were also observed simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18~60 years.
* Serum HBsAg positive.
* Ultrasonographic evidences of cirrhosis.

Exclusion Criteria:

* history of moderate to severe hepatic encephalopathy or variceal bleeding during the last two months before enrolment.
* Prothrombin time is less than 30s.
* Cirrhosis caused by other reasons except HBV infection.
* Severe problems in other vital organs(e.g.the heart,renal or lungs).
* Liver tumor on ultrasonography, CT or MRI examination.
* Pregnant or lactating women.
* Imaging evidences of vascular thromboses.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-10 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
The levels of serum alanine aminotransferase (ALT), total bilirubin (TB),prothrombin time (PT), albumin (ALB), prealbumin(PA), precollagenⅢ(PCⅢ), collagenⅣ(Ⅳ-C), laminin(LN), hyaluronidase(HN), liver histological improvement. | pre-transplantation, and 1week to 1 year post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Lin B liang, MD/PHD, Principal Investigator — SunYat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China